CLINICAL TRIAL: NCT03439748
Title: Reward Sensitivity as a Mechanism of Positive Affect Treatment
Brief Title: Treatment for Affect Dimensions
Acronym: TAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Southern Methodist University (Other)
Responsible Party: Principal Investigator, Michelle Craske, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R61MH115138 (NIH)
Record Dates: First submitted 2018-02-05; First posted 2018-02-20 (Actual); Results first posted 2023-12-07 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Affect Treatment (Experimental): 15 sessions of psychotherapy designed to augment reward anticipation, reward attainment, and reward learning.
  Interventions: Behavioral: Positive Affect Treatment
- Negative Affect Treatment (Active Comparator): 15 sessions of psychotherapy designed to decrease threat avoidance, threat appraisal and arousal.
  Interventions: Behavioral: Negative Affect Treatment

INTERVENTIONS:
Behavioral: Positive Affect Treatment — Sessions 1-7: Pleasurable activities + imaginal recounting and reinforcement of positive mood effects (continued for sessions 8-15) Sessions 8-10: Cognitive exercises focusing on identifying positive aspects of experience, taking responsibility for positive outcomes, and imagining future positive events Sessions 11-14: Exercises to cultivate and savor positive experiences Session 15: Relapse prevention.
  Arms: Positive Affect Treatment
Behavioral: Negative Affect Treatment — Sessions 1-7: Exposure therapy to feared or avoided situations, sensations, or memories (continued for sessions 8-15) Sessions 8-10: Cognitive restructuring of probability, cost, and attributional biases Sessions 11-14: Capnometry-assisted respiratory training Session 15: Relapse prevention
  Arms: Negative Affect Treatment

SUMMARY:
The purpose of this study is to evaluate the efficacy and targets of Positive Affect Treatment, a psychotherapy specifically aimed at enhancing reward sensitivity in individuals with low positive affect (a core feature of anhedonia) in the context of depression or anxiety.

Target enrollment is 68 male and female participants with low positive affect and depression or anxiety and impaired functioning, between the ages of 18 and 65 years, who will be randomized to either Positive Affect Treatment or Negative Affect Treatment (designed to reduce threat sensitivity). Participants will complete laboratory tests, psychiatric assessments, and self-report questionnaires as part of the study.

The total length of participation is around 4 months.

DETAILED DESCRIPTION:
Low positive affect in the context of depression or anxiety has been relatively resistant to pharmacological and psychological treatments. Newer treatments that focus upon positivity or reward sensitivity have shown promising results.

As an NIMH funded R61 phase trial, the purpose of the current randomized controlled trial is to evaluate the efficacy and targets of Positive Affect Treatment (designed to augment reward sensitivity) for individuals with low positive affect in the context of depression or anxiety symptoms. Targets include behavioral, cognitive, physiological and experiential measures of three reward processes: reward anticipation, response to reward attainment, and reward learning. Specificity of target engagement is assessed by comparison with Negative Affect Treatment, designed to reduce threat sensitivity.

Clinical outcomes are assessed at baseline and either weekly or at Week 5, Week 10, and Week 15 (post). Targets are assessed at baseline, Week 5, Week 10, and Week 15. Statistical models evaluate whether change in outcomes and change in target measures are greater as a result of Positive Affect Treatment compared to Negative Affect Treatment and whether changes in target measures correlate with changes in outcome measures.

Target enrollment is 68 male and female participants with low positive affect and depression or anxiety and impaired functioning between the ages of 18 and 65 who will be randomized to Positive Affect Treatment or Negative Affect Treatment, each comprising 15 individual psychotherapy sessions.

Participants will complete laboratory tests and psychiatric assessments and self-report questionnaires as part of the study. Total length of participation is around 4 months.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Low positive affect indexed by less than or equal to 24 on the positive affect subscale of the PANAS (i.e., PANAS-P); and scores of greater than or equal to 11 for depression, greater to or equal to 6 for anxiety, or greater to or equal to 10 for stress on the Depression, Anxiety, and Stress Scale; and scores of greater than or equal to 5 on any Sheehan Disability Scale subscale.
* Willingness to refrain from starting other psychosocial or pharmacological treatments until study completion.

Exclusion Criteria:

* Patient report of serious medical conditions - such as history of serious, uncontrolled medical illness, or instability (including significant cardio-pulmonary disease, organic brain syndrome, seizure disorder, cerebrovascular disease, thyroid dysfunction, and diabetes)
* Active suicidal ideation
* Lifetime history of bipolar disorder, psychosis, mental retardation, or organic brain damage
* Substance abuse in the last 6 months or dependence within last 12 months.
* 11 or more cigarettes per week or nicotine equivalent.
* History of marijuana, cocaine or stimulant use 5-7 times/week or more before age 15 (e.g., amphetamine, cocaine, methamphetamine)
* Pregnancy
* Bupropion, dopaminergic or neuroleptic medication use in the past 6 months
* Heterocyclics and SSRIs are permitted if stabilized (3 months) and PRN benzodiazepines and beta-blockers are permitted but discouraged on laboratory assessment visits
* Refusal of video/audio-taping

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - Southern Methodist University, Dallas, Texas

REFERENCES:
- [Derived] Uribe S, Kumar D, Rosenfield D, Ritz T, Meuret AE. From in-person to virtual: The impact of crisis-enforced delivery change on treatment for low positive affect, depression, and anxiety. J Affect Disord. 2025 Dec 15;391:119864. doi: 10.1016/j.jad.2025.119864. Epub 2025 Jul 11. PMID 40652976
- [Derived] Craske MG, Meuret AE, Echiverri-Cohen A, Rosenfield D, Ritz T. Positive affect treatment targets reward sensitivity: A randomized controlled trial. J Consult Clin Psychol. 2023 Jun;91(6):350-366. doi: 10.1037/ccp0000805. Epub 2023 Mar 9. PMID 36892884

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began February 23, 2019 and ended February 5, 2021. A brief study description was distributed via lab websites, social media, ClinicalTrials.gov, and campus and local area flyers.
Pre-assignment Details: 1062 individuals completed an online screening. 517 were excluded due to ineligibility and 114 did not follow up. 431 were scheduled for a phone screen. 27 declined, 131 were excluded due to ineligibility, and 60 could not be reached. The remaining 213 were scheduled for a diagnostic assessment. 30 declined to participate, 46 were excluded due to ineligibility or other reasons, and 45 could not be reached. 92 participants were eligible. 7 withdrew during or after assessment. 85 were randomized.
Period: Overall Study
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Started | 42 | 43
Week 5 Assessment | 36 | 37
Week 10 Assessment | 32 | 29
Completed | 31 | 26
Not Completed | 11 | 17
Not completed — Withdrawal by Subject | 11 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Affect Treatment | Negative Affect Treatment | Total
Number analyzed (Participants) | 42 | 43 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.95 (11.5) | 31.51 (13.1) | 31.73 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 36 | 67
  Male | 11 | 7 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 28 | 25 | 53
  Asian | 8 | 9 | 17
  Alaska Native/Native American/Indigenous | 1 | 0 | 1
  Pacific Islander/Native Hawaiian | 0 | 1 | 1
  Black or African American | 2 | 3 | 5
  Hispanic/Latino (White) | 6 | 9 | 15
  Hispanic/Latino (non-White) | 4 | 4 | 8
  Multiracial | 3 | 1 | 4
  Other | 1 | 7 | 8
Marital status [Count of Participants; unit: Participants]
  Married | 9 | 10 | 19
  Single, in a relationship | 10 | 13 | 23
  Single, not in a relationship | 19 | 19 | 38
  Separated | 1 | 1 | 2
  Divorced | 3 | 0 | 3
Current psychotropic medication [Count of Participants; unit: Participants] | 12 | 12 | 24
Any diagnosis [Count of Participants; unit: Participants] | 37 | 39 | 76
Depressive diagnoses [Count of Participants; unit: Participants] | 27 | 31 | 58
Major depressive disorder [Count of Participants; unit: Participants] | 19 | 27 | 46
Persistent depressive disorder [Count of Participants; unit: Participants] | 17 | 16 | 33
Anxiety diagnoses [Count of Participants; unit: Participants] | 24 | 26 | 50
Panic disorder [Count of Participants; unit: Participants] | 5 | 5 | 10
Agoraphobia [Count of Participants; unit: Participants] | 1 | 2 | 3
Social anxiety disorder [Count of Participants; unit: Participants] | 17 | 17 | 34
Generalized anxiety disorder [Count of Participants; unit: Participants] | 15 | 16 | 31
Specific phobia [Count of Participants; unit: Participants] | 3 | 4 | 7
Posttraumatic stress disorder [Count of Participants; unit: Participants] | 0 | 3 | 3
Obsessive compulsive disorder [Count of Participants; unit: Participants] | 0 | 3 | 3
Attention deficit hyperactivity [Count of Participants; unit: Participants] | 9 | 5 | 14
Adjustment disorder [Count of Participants; unit: Participants] | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Positive Affect Subscale of the Positive and Negative Affect Scale (PANAS-P)
Description: Reported positive affect. Scores can range from 10-50, with higher scores representing higher levels of positive affect.
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 42 | 43
score on a scale
  Week 0 | 20.76 (7.42) | 29.42 (4.74)
  Week 5: number analyzed (Participants) | 39 | 36
  Week 5 | 24.18 (7.37) | 19.42 (8.12)
  Week 10: number analyzed (Participants) | 33 | 30
  Week 10 | 26.88 (8.29) | 22.57 (9.82)
  Week 16: number analyzed (Participants) | 33 | 26
  Week 16 | 27.30 (7.23) | 23.85 (9.28)
Statistical Analysis 1: Comparison: Positive Affect Treatment vs Negative Affect Treatment; This analysis compares the PAT and NAT groups at post-treatment. For this analysis, we have greater than .80 power to detect an effect size difference between PAT and NAT as small as d=.35; Test type: Superiority; p = .002, Mixed Models Analysis — The threshold for statistical significance was p = 0.05. Univariate tests were corrected for false discovery rate using the Benjamin-Hochberg approach; Baseline levels of outcomes were covaried in all analyses to reduce error variance and correct for group differences

2. Primary Outcome: Interviewer Anhedonia Ratings
Description: Interviewer ratings of interest, pleasure, and motivation in hobbies/pastimes, foods/drinks, social activities (score range: 1-12), higher scores indicate lower anhedonia.
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 42 | 43
score on a scale
  Week 0: number analyzed (Participants) | 41 | 43
  Week 0 | 7.66 (2.13) | 7.47 (1.80)
  Week 5: number analyzed (Participants) | 36 | 37
  Week 5 | 6.11 (2.26) | 5.49 (2.40)
  Week 10: number analyzed (Participants) | 32 | 29
  Week 10 | 4.91 (2.19) | 4.93 (2.40)
  Week 16: number analyzed (Participants) | 32 | 23
  Week 16 | 4.19 (1.47) | 4.43 (2.23)
Statistical Analysis 1: Comparison: Positive Affect Treatment vs Negative Affect Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p > .05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Baseline levels of outcomes were covaried in all analyses to reduce error variance and correct for group differences

3. Primary Outcome: Depression Anxiety and Stress Scale (DASS-21)
Description: Reported symptoms of depression, anxiety, and stress (score range: 0-63), higher scores indicate higher symptom severity and frequency.
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 42 | 43
score on a scale
  Week 0 | 27.36 (11.27) | 24.51 (10.54)
  Week 5: number analyzed (Participants) | 39 | 36
  Week 5 | 17.90 (11.56) | 17.92 (10.51)
  Week 10: number analyzed (Participants) | 33 | 30
  Week 10 | 11.55 (9.60) | 13.00 (12.13)
  Week 16: number analyzed (Participants) | 33 | 26
  Week 16 | 9.09 (6.85) | 12.38 (10.90)
Statistical Analysis 1: Comparison: Positive Affect Treatment vs Negative Affect Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .024, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Baseline levels of outcomes were covaried in all analyses to reduce error variance and correct for group differences

4. Secondary Outcome: Sheehan Disability Scale (SDS)
Description: Reported impairment due to symptoms (score range: 0-30) with higher scores indicating greater impairment. Includes reported number of days of missed school/work and number of days of reduced productivity. Statistical analyses have not yet been conducted for this outcome measure.
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 42 | 43
score on a scale
  Week 0 | 18.40 (6.14) | 16.65 (6.51)
  Week 5: number analyzed (Participants) | 36 | 37
  Week 5 | 14.53 (6.46) | 14.84 (6.97)
  Week 10: number analyzed (Participants) | 32 | 29
  Week 10 | 11.19 (6.34) | 11.86 (6.94)
  Week 16: number analyzed (Participants) | 32 | 26
  Week 16 | 9.56 (6.64) | 9.08 (6.38)

5. Secondary Outcome: Beck Depression Inventory (BDI)
Description: Reported suicidal ideation (item 9 on the BDI), scores range from 0-3 with higher scores indicating a higher degree of suicidal ideation. Statistical analyses have not yet been conducted for this outcome measure.
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 42 | 43
score on a scale
  Week 0 | 0.17 (0.38) | 0.23 (0.43)
  Week 5: number analyzed (Participants) | 39 | 36
  Week 5 | 0.18 (0.39) | 0.14 (0.35)
  Week 10: number analyzed (Participants) | 33 | 30
  Week 10 | 0.18 (0.39) | 0.20 (0.41)
  Week 16: number analyzed (Participants) | 31 | 26
  Week 16 | 0.23 (0.43) | 0.08 (0.27)

6. Secondary Outcome: Daily Activity/Social Interaction (Actigraph)
Description: We intended to collect data on energy expenditure over four 7-day periods (at week 0, week 5, week 10, and week 16) using a wrist-worn Actigraph tri-axial accelerometer. However, the use of Actigraph monitors was terminated early in the study due to the onset of the COVID-19 pandemic.
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: kcals expended per hour
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 15 | 14
kcals expended per hour
  Week 0 | 40.212 (19.677) | 34.634 (24.427)
  Week 5 | 41.98 (20.58) | 41.44 (26.06)
  Week 10 | 34.21 (20.75) | 46.92 (29.33)
  Week 16 | 43.69 (27.13) | 56.57 (53.04)

7. Secondary Outcome: Effort Expenditure for Rewards Task (EEfRT)
Description: The Effort Expenditure for Rewards Task (EEfRT) is a computer-based multi-trial task used to objectively assess decision-making and willingness to expend effort for reward. The dependent variable is the ratio of hard (high-effort) choices to the total number of trials. Results range from 0 to 1, with higher values indicating a higher proportion of hard (high-effort) choices. Results show the mean proportion of high-effort choices.
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: proportion of high effort choices
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 42 | 43
proportion of high effort choices
  Week 0: number analyzed (Participants) | 27 | 22
  Week 0 | 0.41 (0.20) | 0.41 (0.27)
  Week 5: number analyzed (Participants) | 24 | 23
  Week 5 | 0.43 (0.22) | 0.39 (0.23)
  Week 10: number analyzed (Participants) | 19 | 12
  Week 10 | 0.51 (0.26) | 0.41 (0.31)
  Week 16: number analyzed (Participants) | 18 | 12
  Week 16 | 0.48 (0.29) | 0.42 (0.32)
Statistical Analysis 1: Comparison: Positive Affect Treatment vs Negative Affect Treatment; This analysis compares the PAT and NAT groups at post-treatment. For this analysis, we have greater than .80 power to detect an effect size difference as small as d=.39; Test type: Superiority; p = .922, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Baseline levels of outcomes were covaried in all analyses to reduce error variance and correct for group differences

8. Secondary Outcome: Monetary Incentive Task
Description: Heart rate acceleration during the Monetary Incentive Task (MIT) was used to measure cardiac responding to the prospect of a monetary reward. The dependent variable is the interbeat interval acceleration during the task (score range in our sample: -0.16 to 0.17). Higher values indicate greater cardiac responding to the prospect of monetary reward.
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: beats/ms^2
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 42 | 43
beats/ms^2
  Week 0: number analyzed (Participants) | 34 | 38
  Week 0 | -0.012 (0.512) | -0.017 (0.046)
  Week 5: number analyzed (Participants) | 24 | 29
  Week 5 | 0.017 (0.048) | 0.013 (0.061)
  Week 10: number analyzed (Participants) | 19 | 18
  Week 10 | -0.002 (0.042) | 0.004 (0.043)
  Week 16: number analyzed (Participants) | 16 | 13
  Week 16 | 0.003 (0.026) | 0.026 (0.053)
Statistical Analysis 1: Comparison: Positive Affect Treatment vs Negative Affect Treatment; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = .049, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Baseline levels of outcomes were covaried in all analyses to reduce error variance and correct for group differences

9. Secondary Outcome: Behavioral Inhibition/Behavioral Activation (Reward Drive Subscale) (BAS-RD)
Description: Mediator: Reported reward sensitivity (score range: 4-16), with higher scores indicating higher sensitivity
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 42 | 43
score on a scale
  Week 0 | 9.67 (2.63) | 9.42 (2.21)
  Week 5: number analyzed (Participants) | 36 | 37
  Week 5 | 10.50 (2.63) | 10.14 (2.26)
  Week 10: number analyzed (Participants) | 32 | 29
  Week 10 | 10.66 (2.51) | 10.66 (2.36)
  Week 16: number analyzed (Participants) | 33 | 26
  Week 16 | 10.30 (2.56) | 11.08 (1.96)
Statistical Analysis 1: Comparison: Positive Affect Treatment vs Negative Affect Treatment; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = .591, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Baseline levels of outcomes were covaried in all analyses to reduce error variance and correct for group differences

10. Secondary Outcome: Dimensional Anhedonia Rating Scale-Anticipation and Motivation Items
Description: Mediator: Reported reward desire, motivation, and effort (score range: 0-76) with higher scores indicating higher degree of reward desire, motivation, and effort.
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 42 | 43
score on a scale
  Week 0: number analyzed (Participants) | 41 | 43
  Week 0 | 42.85 (16.96) | 49.16 (16.32)
  Week 5: number analyzed (Participants) | 36 | 37
  Week 5 | 52.28 (14.20) | 52.46 (15.36)
  Week 10: number analyzed (Participants) | 32 | 29
  Week 10 | 55.63 (15.69) | 55.66 (16.08)
  Week 16: number analyzed (Participants) | 32 | 26
  Week 16 | 59.84 (14.31) | 58.46 (16.31)
Statistical Analysis 1: Comparison: Positive Affect Treatment vs Negative Affect Treatment; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = .004, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Baseline levels of outcomes were covaried in all analyses to reduce error variance and correct for group differences

11. Secondary Outcome: Dimensional Anhedonia Rating Scale-Consummatory Items
Description: Mediator: Reported reward-related pleasure (score range: 0-28), with higher scores indicating higher degree of pleasure.
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 42 | 43
score on a scale
  Week 0: number analyzed (Participants) | 41 | 43
  Week 0 | 17.56 (6.26) | 19.12 (6.16)
  Week 5: number analyzed (Participants) | 36 | 37
  Week 5 | 20.39 (4.76) | 20.51 (6.25)
  Week 10: number analyzed (Participants) | 32 | 29
  Week 10 | 21.50 (5.66) | 21.59 (5.99)
  Week 16: number analyzed (Participants) | 32 | 26
  Week 16 | 22.88 (4.73) | 22.12 (5.78)
Statistical Analysis 1: Comparison: Positive Affect Treatment vs Negative Affect Treatment; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = .030, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Baseline levels of outcomes were covaried in all analyses to reduce error variance and correct for group differences

12. Secondary Outcome: Modified Attentional Dot Probe Task-Disengagement Bias for Negative Stimuli
Description: The Modified Attentional Dot Probe Task is a computer-based multi-trial task used to objectively assess attentional bias toward positively- and negatively-valenced stimuli. The dependent variable is the reaction time index for disengagement bias from sad faces. This is calculated as follows: (Cue appears proximal to emotional face in the pair of emotional face and random blur image: reaction time for target distal to emotional face minus reaction time for target proximal to emotional face) minus (Cue proximal to neutral face in pair of neutral face and random blur image: reaction time for target distal to neutral face minus reaction time for target proximal to neutral face). The range of values in our sample was: -309.28 to 283.45.
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 42 | 43
milliseconds (ms)
  Week 0: number analyzed (Participants) | 36 | 38
  Week 0 | -43.43 (114.62) | 2.80 (105.63)
  Week 5: number analyzed (Participants) | 26 | 29
  Week 5 | 16.70 (98.11) | -16.49 (102.44)
  Week 10: number analyzed (Participants) | 21 | 18
  Week 10 | -3.07 (82.01) | -31.56 (94.05)
  Week 16: number analyzed (Participants) | 19 | 14
  Week 16 | 4.85 (97.00) | 66.24 (101.47)
Statistical Analysis 1: Comparison: Positive Affect Treatment vs Negative Affect Treatment; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = .029, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

13. Secondary Outcome: Modified Attentional Dot Probe Task-Engagement Bias for Positive Stimuli
Description: The Modified Attentional Dot Probe Task is a computer-based multi-trial task used to objectively assess attentional bias toward positively- and negatively-valenced stimuli. The dependent variable is the reaction time index for engagement bias from happy faces. This is calculated as follows: (Cue probe distal to negative image in negative/abstract image pair: RT for target probe distal to negative image minus RT for target probe proximal to negative image) minus (Cue probe distal to neutral image in neutral/abstract image pair: RT for target probe distal to neutral image minus RT for target probe proximal to neutral image). The range of data in our sample was: -237.82 to to 343.93. Statistical analyses have not yet been conducted for this outcome measure.
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 42 | 43
milliseconds (ms)
  Week 0: number analyzed (Participants) | 36 | 38
  Week 0 | 9.30 (105.87) | 3.29 (108.57)
  Week 5: number analyzed (Participants) | 26 | 29
  Week 5 | -17.65 (90.72) | 2.62 (96.57)
  Week 10: number analyzed (Participants) | 21 | 18
  Week 10 | -20.86 (69.89) | -22.51 (88.93)
  Week 16: number analyzed (Participants) | 19 | 14
  Week 16 | -22.51 (89.93) | 16.36 (111.56)

14. Secondary Outcome: International Affective Picture System Task
Description: Heart rate acceleration during presentation of images from the International Affective Picture Systems (IAPS) was used to assess cardiac responding to positive images. The dependent variable is heart rate acceleration during the 6 seconds of positive image presentation relative to the last 2 seconds before picture onset. Higher values indicate greater cardiac responding to positive images. The range of values in our sample was: -0.12 to 0.09.
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: beats/ms^2
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 42 | 43
beats/ms^2
  Week 0: number analyzed (Participants) | 30 | 37
  Week 0 | 0.0003 (0.0243) | -0.0007 (0.0238)
  Week 5: number analyzed (Participants) | 25 | 28
  Week 5 | -0.0016 (0.0222) | -0.0061 (0.0331)
  Week 10: number analyzed (Participants) | 20 | 19
  Week 10 | 0.0071 (0.0221) | 0.0013 (0.0244)
  Week 16: number analyzed (Participants) | 20 | 13
  Week 16 | 0.0024 (0.0222) | 0.0035 (0.0524)
Statistical Analysis 1: Comparison: Positive Affect Treatment vs Negative Affect Treatment; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = .494, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Baseline levels of outcomes were covaried in all analyses to reduce error variance and correct for group differences

15. Secondary Outcome: Temporal Experience of Pleasure Scale (Consummatory Subscale)
Description: Mediator: Reported reward consummatory pleasure (score range: 8-48), with higher scores indicating higher reported reward consummatory pleasure
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 42 | 43
score on a scale
  Week 0 | 35.81 (6.98) | 37.12 (6.03)
  Week 5: number analyzed (Participants) | 36 | 37
  Week 5 | 36.28 (6.20) | 37.49 (5.83)
  Week 10: number analyzed (Participants) | 32 | 29
  Week 10 | 37.03 (6.17) | 37.97 (5.17)
  Week 16: number analyzed (Participants) | 33 | 26
  Week 16 | 37.70 (4.73) | 37.62 (5.59)
Statistical Analysis 1: Comparison: Positive Affect Treatment vs Negative Affect Treatment; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = .231, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Baseline levels of outcomes were covaried in all analyses to reduce error variance and correct for group differences

16. Secondary Outcome: Probabilistic Reward Task (PRT)
Description: The Probabilistic Reward Task (PRT) is a computer-based multi-trial task used to objectively assess the propensity to modulate behavior as a function of prior reinforcements. The dependent variable is response bias (measured as accuracy) toward the more frequently rewarded stimulus. A high response bias emerges when subjects show high rates of correct identification (hits) for the rich stimulus and high miss rates for the lean stimulus (i.e., the stimulus associated with less frequent rewards). Higher values indicate a greater propensity to modulate behavior as a function of prior reinforcements. The range of values in our sample was: -0.58 to 0.78.
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 42 | 43
Ratio
  Week 0: number analyzed (Participants) | 35 | 37
  Week 0 | 0.16 (0.19) | 0.15 (0.29)
  Week 5: number analyzed (Participants) | 27 | 29
  Week 5 | 0.04 (0.27) | 0.19 (0.27)
  Week 10: number analyzed (Participants) | 21 | 18
  Week 10 | 0.09 (0.13) | 0.03 (0.18)
  Week 16: number analyzed (Participants) | 18 | 14
  Week 16 | 0.16 (0.21) | 0.15 (0.23)
Statistical Analysis 1: Comparison: Positive Affect Treatment vs Negative Affect Treatment; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = .344, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Baseline levels of outcomes were covaried in all analyses to reduce error variance and correct for group differences

17. Secondary Outcome: Pavlovian Instrumental Transfer Task - Force (PIT-FORCE)
Description: The Pavlovian Instrumental Transfer (PIT) task assesses the extent to which a conditional stimulus paired with reward influences instrumental responding to gain rewards. The dependent variable was handgrip force exerted in response to stimuli during a test phase following Pavlovian conditioning. Higher values indicate greater instrumental responding to gain rewards as a function of Pavlovian conditioning to a conditional stimulus paired with reward. The range of values in our sample was: -18.76 to 61.30.
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: volts
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 42 | 43
volts
  Week 0: number analyzed (Participants) | 31 | 32
  Week 0 | 6.30 (12.29) | 4.91 (13.54)
  Week 5: number analyzed (Participants) | 20 | 21
  Week 5 | 7.96 (15.61) | 6.72 (12.60)
  Week 10: number analyzed (Participants) | 16 | 13
  Week 10 | 6.55 (16.39) | 6.57 (12.35)
  Week 16: number analyzed (Participants) | 11 | 8
  Week 16 | 8.05 (16.34) | 1.24 (7.96)
Statistical Analysis 1: Comparison: Positive Affect Treatment vs Negative Affect Treatment; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = .267, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Baseline levels of outcomes were covaried in all analyses to reduce error variance and correct for group differences

18. Secondary Outcome: Pavlovian Instrumental Transfer Task - Valence (PIT-VALENCE)
Description: Within the Pavlovian Instrumental Transfer Task (PIT), participants rate the pleasantness (0-4) for three conditional stimuli to indicate the perceived value of reward associated with each one. The dependent variable is the self-reported pleasantness for rewarded stimuli compared to nonrewarded stimuli. This is calculated by first taking the average of participants' pleasantness ratings for the three CS+s and CS-s, and then subtracting the average CS- ratings from the average CS+ ratings. Higher values indicate greater responding to Pavlovian conditioning during the task.
Time Frame: Week 0, Week 5, Week 10, Week 16
Population: Intent to treat population (all participants assigned to Positive Affect Treatment or Negative Affect Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
Number analyzed (Participants) | 42 | 43
score on a scale
  Week 0: number analyzed (Participants) | 32 | 43
  Week 0 | 1.09 (2.10) | 0.62 (2.17)
  Week 5: number analyzed (Participants) | 22 | 26
  Week 5 | 1.50 (2.50) | 0.73 (2.99)
  Week 10: number analyzed (Participants) | 21 | 18
  Week 10 | 1.29 (2.88) | 0.44 (2.94)
  Week 16: number analyzed (Participants) | 19 | 14
  Week 16 | 0.74 (2.49) | 1.93 (1.90)
Statistical Analysis 1: Comparison: Positive Affect Treatment vs Negative Affect Treatment; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = .051, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Baseline levels of outcomes were covaried in all analyses to reduce error variance and correct for group differences

ADVERSE EVENTS:
Time Frame: Each participant was assessed over 16 weeks
Description: DSMB committee members independently evaluated whether each event qualified as a serious adverse event using the following criteria: 1) Serious/Not serious: Is the event serious or places subjects or others at greater risk than previously known or recognized? 2) Expected/Unexpected: Is the event unexpected (not described in the protocol or consent or exceeds severity/frequency of expected event) 3) Causality: Is the event-related or possibly related to research procedures?
Arm/Group | Positive Affect Treatment | Negative Affect Treatment
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/43
Other Adverse Events (participants affected / at risk) | 0/42 | 3/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Positive Affect Treatment (N=42) | Negative Affect Treatment (N=43)
Clinical deterioration (Psychiatric disorders) | 0 (0) | 2 (2) — Two participants experienced clinical deterioration during treatment. For both, the team decided that the participant's therapist would go off-protocol following session 10 in order to best address the participant's current mental health needs.
Homework noncompliance leading to participant withdrawal (Psychiatric disorders) | 0 (0) | 1 (1) — Participant did not complete homework for NAT sessions 5-11. Participant also expressed ambivalence about completing CART protocol between sessions. Following introduction of CART protocol, they expressed that they would like to terminate services.

LIMITATIONS AND CAVEATS:
Generalizability from academic to community settings; Sample was selected to have low positive affect, thus results may not generalize to samples diagnosed with anhedonia; Lack of follow-up assessment prevented evaluation of long-term changes in target measures and outcomes; Sample powered for moderate or larger effects, while smaller effects may require larger samples; Participants not blinded to condition; NAT was not representative of typical cognitive-behavioral therapy for depression.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/48/NCT03439748/Prot_SAP_ICF_000.pdf